CLINICAL TRIAL: NCT02334241
Title: The Sorbact® Antimicrobial Dressing in the Holistic Wound Management Of Diabetic Foot ulCers (Phase III Study)
Acronym: ADHOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INRESA Pharma (Industry)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INR 2014-001
Record Dates: First submitted 2014-12-11; First posted 2015-01-08 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Sorbact; Best local Cares; DFU
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorbact® (Experimental): The basic Sorbact® presentation is an antimicrobial, non-adhesive absorbent wound dressing. It consists of a highly absorbent hydropolymer matrix with an antimicrobial Sorbact® mesh (Sorbact® acetate fabric coated with dialkyl carbamoyl chloride - DACC) and is covered by a semipermeable polyurethane film.
  Interventions: Device: Sorbact®
- Best local cares (Active Comparator): Dressing requirements in this study have to be consistent with international guidelines.
  Interventions: Device: Best local cares

INTERVENTIONS:
Device: Sorbact® — Sorbact® is available in many types and sizes. These different presentations are available allowing management of quite all types of wounds of various anatomical locations, sizes or depths. Application of any of these presentations is allowed and may change during study course according to wound evolution.
  Arms: Sorbact®
Device: Best local cares — Participating centers will provide a list of dressings they planned to use in the best local cares arm. This list must be validated by the study Steering Committee members
  Arms: Best local cares

SUMMARY:
The aim of this study is to demonstrate, during a 12-week follow-up, a greater efficacy of using Sorbact® dressing technology in addition to best local cares compared to best local cares alone in the management of diabetic foot ulcers

DETAILED DESCRIPTION:
This study will select a target population of diabetic patients treated for foot ulcers of neuropathic origin, with or without arterial disease but not presenting critical limb ischaemia. No definitive wound infection should be present at inclusion. According to randomization, all present ulcers at baseline will be treated either with best local cares not including Sorbact® dressing or including systematically for all ulcers this medical device.

The main study endpoint will be a composite criterion defining a favourable limb outcome for a given patient. This criterion will be considered as present if total open wound area has decreased by 50% or more at last available evaluation whereas no definitive infection has occurred and no amputation has been required.

Patients will be followed over a maximal period of 12 weeks. At D0 (inclusion), W2, W4, W6, W8, W10 and W12 a detailed description of ulcer aspect will be done. Applied dressing will be removed according to a standardized procedure. Wound area tracing and photography of all ulcers will be performed. Off-loading system's adherence will be checked.

Between these weekly evaluations, all performed local cares will be reported and each dressing removal will be performed by using a similar procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent to participate obtained.
2. Male or female patient aged at least 18 years without superior limit.
3. Type 1 or 2 diabetes.
4. Less than one month HbA1c <=10%.
5. Presence, on at least one foot, of a full-thickness ulcer for at least 4 weeks (location below the malleola).
6. Neuropathy confirmed by insensitivity to monofilament (Semmes-Weinstein 5.07 monofilament according to diagnosis criteria presented in appendix 05).
7. No ulcer should present a moderate or severe infection at baseline. Concomitant treatment with systemic antibiotics at baseline is accepted if all ulcers meet none of the criteria defining moderate or severe infection.
8. All ulcers are appropriately debrided (less than 10% black tissue covering wound area on a colorimetric scale, adequate removal of hyperkeratosis).
9. All ulcers are of Grade 1 or 2 of the Wagner classification.
10. Ulcers should meet one of the following criteria:

    If only one ulcer is present, its largest diameters has to be ≥1 cm or this ulcer is categorized as grade 2 according to Wagner classification If more than one ulcer is present, the sum of all largest diameters has to be ≥2 cm or one ulcer is categorized as grade 2 according to Wagner classification
11. For both legs: ABPI ≥0.6 and <1.3 AND ankle systolic pressure ≥70 mmHg or systolic toe pressure ≥50 mmHg or TcPo2 ≥30 mmHg (decubitus).

    If ABPI ≥1.3, patent femoral artery inflow should be confirmed by digital angiography, magnetic resonance, or CT angiography or doppler ultrasonography <6 months before randomization.
12. Patient compliant to one of the accepted off-loading system.

Exclusion Criteria:

1. Previous history of major amputation (cf. § 10.3.3.2 for definition) or planned major amputation within the first month after randomization.
2. Revascularization procedure of lower leg, or any other treatment (e.g. neurostimulation) of any leg <8 weeks before randomization.
3. Patient unable to be treated with one of the accepted type of off-loading system.
4. Active Charcot foot.
5. Presence of any ulcer with evidence of skin cancer.
6. Presence of another chronic wound (i.e. present for 4 weeks or more) not involving the foot or involving the foot but extending above malleolus.
7. Patient suffering from any known active malignancy, other than basal-cell carcinoma and cervical carcinoma in situ, requiring any general, local, surgical or radiation therapy.
8. Patient suffering from severe morbid obesity (BMI ≥50 kg/m2).
9. Severe hypertension with systolic blood pressure ≥180 mm Hg or diastolic blood pressure ≥110 mm Hg (measured at two occasions separated by a 4 week period in a patient sitting for at least 5 min).
10. Patient with a severe comorbid disorder, not expected to survive more than 12 months
11. Acute cardiovascular events (e.g. myocardial infarction, stroke, recent coronary intervention) within 3 months before randomisation
12. Patient who are in the exclusion period following a previous participation to another trial or who are currently participating to any concomitant study with any drug or device.
13. Known intolerance to the tested medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Favourable healing outcome (FHO) | 12 weeks
  A FHO is considered to have occurred in a given patient if all the following composite endpoints are met:
  I. Total wound area (sum of areas of all present wounds on both limbs) has decreased, compared to baseline, by 50% or more at last available evaluation.
  II. No minor or major amputation decided during the follow-up period. III. No moderate/severe infection of any present wound has been detected during the follow-up period.

SECONDARY OUTCOMES:
Comparative evaluation of each of the items used to define a FHO. | 12 weeks
Time to reach a 50% total wound area reduction. | 12 weeks
Comparative evaluation of the number of complete wound closure. | 12 weeks
Comparative evaluation of total absolute and relative wound area regression and of total wound edge migration (Gilman's formula; sum of the score of each individual ulcer) over 12 weeks (centralized analysis of wound area tracings). | 12 weeks
Number of local cares requiring instrumental debridement (surgical or sharp debridement). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan APELQVIST, Principal Investigator — University Hospital of Malmö
Locations (15):
- Czechia (5):
  - Faculty of Medicine MU a FH St. Ann Brno, Brno
  - Cardiologic and pediatric ambulance s.r.o., Ostrava-vitkovice
  - Institute for Clinical and Experimental Medicine, Prague
  - Podiatrie - Ustredni vojenska nemocnice - Vojenska fakultni nemocnice Praha, Prague
  - Bulovka Hospital, Prague
- France (5):
  - Hôpital Cardio-vasculaire Louis Pradel, Bron
  - CHRU LILLE Hôpital Claude Huriez, Lille
  - CHRU Lapeyronie, Montpellier
  - Hopital Civil, Strasbourg
  - Maison de santé protestante de Bordeaux Bagatelle, Talence
- Poland (5):
  - Gdański Uniwersytet Medyczny, Gdansk
  - Instytut Medycny Wsi, Lublin
  - Angiodiabetica, Poznan
  - Warszawski Uniwersytet Medyczny, Warsaw
  - PODOS, Warsaw